CLINICAL TRIAL: NCT00536497
Title: A 2 Part Open-label, Randomised, Crossover Study to Compare the Effects of Formulation, Food and Particle Size on the Pharmacokinetic Profiles of a Single 175mg Dose of GW842166X in Healthy Male and Female Volunteers
Brief Title: Relative Bioavailability Study on a Single Dose of GW842166X in Healthy Male and Female Subjects.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Compound terminated
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CBA109358
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Subjects
Keywords: GW842166,; Healthy volunteers,; Inflammatory Pain.
MeSH Terms: interventions — 2-((2,4-dichlorphenyl)amino)-N-((tetrahydro-2H-pyran-4-yl)methyl)-4-(trifluoromethyl)-5-pyrimidinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW842166X

SUMMARY:
GW842166X is a selective non-cannabinoid CB2 receptor agonist, which is undergoing clinical development as a novel oral treatment for inflammatory pain. The purpose of the study is to compare the effects of formulation, food and particle size on the pharmacokinetic profiles of a single 175mg dose of GW842166X in healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >50 Kg and BMI within the range 18.5-29.9 Kg/m2 inclusive.
* Healthy as judged by a responsible physician.

Exclusion Criteria:

* Positive pre-study urine screen for drugs of abuse or alcohol breath test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Plasma GW842166 Cmax and AUC (O-Infinity) | Timepoints: Pre dose, 15 mins, 30 mins, 45 mins, 1hr, 1.5hrs, 2hrs, 2.5hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, 12hrs, 16hrs, 24hrs, 48hrs, 48hr, 96hrs (post dose)

SECONDARY OUTCOMES:
Plasma GW842166 AUC (0-t), tlag,tmax and t1/2 | Timepoints: Pre dose, 15 mins, 30 mins, 45 mins, 1hr, 1.5hrs, 2hrs, 2.5hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, 12hrs, 16hrs, 24hrs, 48hrs, 48hr, 96hrs (post dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline